CLINICAL TRIAL: NCT02129959
Title: Cardiovascular Effects of the Degree of Head-down and Pneumoperitoneum During Laparoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, VS, National Taiwan University Hospital
Other Study IDs: 201401041RINC
Record Dates: First submitted 2014-05-01; First posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Laparoscopy
Keywords: laparoscopic cholecystectomy, laparoscopic gastrectomy, laparoscopic colectomy, laparoscopic appendectomy, laparoscopic; assisted vaginal hysterectomy, robot-assisted laparoscopic radical prostatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- laparoscopy: laparoscopic cholecystectomy, laparoscopic gastrectomy, laparoscopic colectomy, laparoscopic appendectomy, laparoscopic assisted vaginal hysterectomy, robot-assisted laparoscopic radical prostatectomy

SUMMARY:
The aim of this study is to observe the cardiovascular effects of the degree of head-down angle and pneumoperitoneum during laparoscopic procedure using by the fourth version Vigileo-Flotrac system.

DETAILED DESCRIPTION:
Laparoscopy for general surgery followed and proved to be advantageous in reduction of postoperative pain, better cosmetic results, quicker return to normal activities, reduction in hospital stay resulting in overall reduction in medical cost, less intraoperative bleeding, less postoperative pulmonary complications, less postoperative wound infection, reduced metabolic derangement, and better postoperative respiratory function. In recent years, advanced laparoscopic surgery has targeted older and sicker patients, rendering anesthesia during laparoscopy more technically demanding. Robotic-assisted laparoscopic radical prostatectomy is rapidly becoming a part of the standard surgical repertoire for the treatment of prostate cancer. Robotic-assisted laparoscopic radical prostatectomy are primarily related to the use of pneumoperitoneum in the steep Trendelenburg position. This combination will affect cerebrovascular, respiratory and hemodynamic homeostasis. The golden standard method for measuring cardiac output in the clinical setting is thermodilution using a pulmonary artery catheter, but the risk of pulmonary artery catheter insertion can not be justified in routine cases. The Vigileo-FloTrac system (Edwards Lifesciences, Irvine, CA, USA), is a less invasive method to obtain continuous CO using pulse contour analysis. The aim of this study is to observe the cardiovascular effects of the degree of head-down angle and pneumoperitoneum during laparoscopic procedure using by the fourth version Vigileo-Flotrac system.

We choose 180 ASA physical status I to III patients undergoing laparoscopic surgery are enrolled in this study. These surgical procedures include laparoscopic cholecystectomy, laparoscopic gastrectomy, laparoscopic colectomy, laparoscopic appendectomy, laparoscopic assisted vaginal hysterectomy, robot-assisted laparoscopic radical prostatectomy. These surgical procedures provide the information about the different degree of head-down angle and different intra-abdominal pressure of pneumoperitoneum. Hemodynamic data are recorded immediately after induction of anesthesia; 5 min after induction of pneumoperitoneum; 5, 15, 30, 60 min, and every 30 min if duration more than 60 min after placement in the Trendelenburg position with pneumoperitoneum; and the end.

After observing the cardiovascular effects of degree of head-down, insufflation pressure, duration of surgery, we can prevent the possible complications in advance during laparoscopic surgery. After completing the study, we will be familiar with the use of Vigileo-FloTrac system. We will have more experiences to deal with high-risk patients undergoing simple surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I to III patients undergoing laparoscopic surgery are enrolled in this study.

Exclusion Criteria:

* preoperative ECG reports and severe obesity (body mass index ≥35 kg/m2)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 180 ASA physical status I to III patients undergoing laparoscopic surgery are enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
cardiovascular effects | one year
  Hemodynamic data are recorded immediately after induction of anesthesia; 5 min after induction of pneumoperitoneum; 5, 15, 30, 60 min, and every 30 min if duration more than 60 min after placement in the Trendelenburg position with pneumoperitoneum; and the end.

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH, Taipei, Taiwan, Taiwan